CLINICAL TRIAL: NCT02083666
Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of SOBI002 Following Subcutaneous and Intravenous Administration. A Double-blind, Placebo-controlled, Randomized Within Dose Cohort, Single and Repeated Dose-escalation Study in Healthy Volunteers
Brief Title: Safety and Tolerability of SOBI002 in Healthy Volunteers Following Single and Repeated Administration
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Transient adverse events observed
Sponsor: Swedish Orphan Biovitrum (Industry)
Collaborators: Richmond Pharmacology Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SOBI002-001
Record Dates: First submitted 2014-01-15; First posted 2014-03-11 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Healthy
Keywords: Phase I; Dose cohorts; Escalating dose; Single dose; Multiple dose; Safety; Tolerability; Pharmacokinetics; Pharmacodynamics; volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- SOBI002 (Experimental): Single and repeated administration of different doses of test product
  Interventions: Drug: SOBI002
- placebo (Placebo Comparator): Single and repeated administration of placebo comparator
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SOBI002 — Test Product
  Arms: SOBI002
Drug: Placebo — Reference product
  Arms: placebo

SUMMARY:
The main purpose of this study is to assess the safety and tolerability of SOBI002 in healthy volunteers following single and repeated administration.

DETAILED DESCRIPTION:
This is a double-blind, placebo-controlled, randomized within dose cohort single and repeated dose study with sequential dose escalation.

Eligible volunteers will be divided into dose cohorts and for each cohort, a new panel of 8 volunteers will be randomized to receive either SOBI002 (n=6) or placebo (n=2). SOBI002 will either be administered subcutaneously or intravenously.

ELIGIBILITY:
Inclusion Criteria:

* Females of non-childbearing potential or males
* 18 to 45 years of age
* Judged by the Principal Investigator to be healthy on the basis of medical history and a pre-study physical examination including 12-lead electrocardiogram (ECG), 24-hour Holter ECG, vital signs and blood and urine laboratory assessments.

Exclusion Criteria:

* Females of childbearing potential
* Clinically significant disease
* Clinically significant abnormal laboratory, ECG, vital signs or other safety findings as determined by medical history, physical examination or other evaluations conducted at screening or on admission.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2013-12; Primary Completion 2014-11 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of SOBI002 in healthy volunteers following single and repeated adminstration | Up to 13 weeks
  Safety will be evaluated by assessing all Adverse Events, vital signs, 12-lead ECGs, urine samples for determination of urinalysis variables and blood samples for determination of hematology, biochemistry and coagulation variables.

SECONDARY OUTCOMES:
Assessment of pharmacokinetics of SOBI002 through analysis of serum samples | Up to 13 weeks
Assessment of pharmacodynamics by assessing the inhibition of SOBI002 on hemolytic activity | Up to 13 weeks
Assessment of the immungenicity of SOBI002 by measuring the occurence of anti-drug antibodies | Up to 13 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Erik Brouwer, MD, Study Director — Swedish Orphan Biovitrum AB (publ)
Locations (1):
- Richmond Pharmacology Ltd., London, Saint George's University of London, United Kingdom